CLINICAL TRIAL: NCT04090840
Title: Lifestyle Intervention Feasibility for Arrhythmia and Symptoms With Intermittent Fasting (LIFE AS IF)
Acronym: LIFE AS IF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB19-0879
Record Dates: First submitted 2019-09-11; First posted 2019-09-16 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Obesity; Morbid Obesity; Diabetes Mellitus, Type 2; Atrial Fibrillation
Keywords: obesity; fasting; diet
MeSH Terms: conditions — Obesity; Obesity, Morbid; Diabetes Mellitus, Type 2; Atrial Fibrillation; Fasting

STUDY DESIGN:
Intervention Model Description: Prospective observation study of lifestyle intervention with intermittent fasting (time-restricted eating) of 16 hours every day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intermittent Fasting (Experimental): Patients will follow intermittent fasting for 16 hours with time restricted eating during an 8 hour window. The subjects are also advised to minimize sugar intake to <15g per serving.
  Interventions: Behavioral: Intermittent Fasting

INTERVENTIONS:
Behavioral: Intermittent Fasting — Time restricted eating for 8 hours per day, with 16 hour fast. During the daily fast, patients are encouraged to drink water, black coffee, or green tea without sugar, cream, milk, or sweeteners.

SUMMARY:
BACKGROUND AND RATIONALE

Two out of three Americans are overweight and obesity is associated with hypertension, sleep apnea, atrial fibrillation. Metabolic syndrome with centripetal obesity is also a precursor to insulin resistance and the development of Type II diabetes mellitus. While multiple strategies for weight reduction are often recommended in physician visits, calculating calories and energy expenditure is often inconvenient and does not promote compliance. Intermittent fasting, or time-restricted eating, is a methods to limit caloric intake by fasting for 16 hours to promote ketosis and suppress insulin secretion. Weight loss and reduction in body fat has been observed with brief periods of intervention as time-restricted eating results in reduction in overall caloric intake. Prospective feasibility studies and randomized comparative trials with intermittent fasting are lacking.

The investigators recommend caloric restriction in all of our patients that suffer from arrhythmias and BMI >30. However, they have not systematically measured compliance and the efficacy of lifestyle interventions. Lifestyle counseling and weight loss has been shown to decrease the progression and burden of symptomatic atrial fibrillation. Intermittent fasting can result in consistent reductions in body fat and weight without specific lifestyle counseling. The aim of the present observation cohort study is to assess the feasibility of recommending intermittent fasting in an arrhythmia clinic with regard to compliance and efficacy.

The investigators hypothesize that compliance and adherence to a 16/8 intermittent fasting regimen will be >25% and result in weight loss, compared to the 6 month trend prior to the intervention. This pilot study will serve as the basis to power the first randomized trial comparing intermittent fasting with other types of dietary counseling for arrhythmia outcomes.

OBJECTIVES

To prospectively assess compliance to prescribed intermittent fasting, measured by adherence and change in weight at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* BMI≥ 30
* Ongoing evaluation and management of cardiac arrhythmias

Exclusion Criteria:

* Pregnant or nursing
* Eating disorder or history of eating disorders (self-report)
* Diabetic mellitus type 1 or insulin requiring type 2 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Weight loss | 6 months
  Patients will be weighed weekly for the first month and than have weight checks in clinic monthly

SECONDARY OUTCOMES:
Body Mass Index | Monthly until 6 months
  calculated from height and weight measured in clinic
Waist Circumference | Monthly until 6 months
  measured by research specialist at umbilicus
Blood Pressure | Monthly until 6 months
  measured in clinic by nursing staff
Quality of Life Assessment | 6 months
  SF36 Questionnaire to be filled out by patient
Hemoglobin a1c | 6 months
  Blood test in patients with diabetes mellitus

CONTACTS AND LOCATIONS:
Overall Officials: Roderick Tung, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnosky AR, Hoddy KK, Unterman TG, Varady KA. Intermittent fasting vs daily calorie restriction for type 2 diabetes prevention: a review of human findings. Transl Res. 2014 Oct;164(4):302-11. doi: 10.1016/j.trsl.2014.05.013. Epub 2014 Jun 12. PMID 24993615
- [Background] Moro T, Tinsley G, Bianco A, Marcolin G, Pacelli QF, Battaglia G, Palma A, Gentil P, Neri M, Paoli A. Effects of eight weeks of time-restricted feeding (16/8) on basal metabolism, maximal strength, body composition, inflammation, and cardiovascular risk factors in resistance-trained males. J Transl Med. 2016 Oct 13;14(1):290. doi: 10.1186/s12967-016-1044-0. PMID 27737674
- [Background] Horne BD, Muhlestein JB, Anderson JL. Health effects of intermittent fasting: hormesis or harm? A systematic review. Am J Clin Nutr. 2015 Aug;102(2):464-70. doi: 10.3945/ajcn.115.109553. Epub 2015 Jul 1. PMID 26135345
- [Background] Abed HS, Wittert GA, Leong DP, Shirazi MG, Bahrami B, Middeldorp ME, Lorimer MF, Lau DH, Antic NA, Brooks AG, Abhayaratna WP, Kalman JM, Sanders P. Effect of weight reduction and cardiometabolic risk factor management on symptom burden and severity in patients with atrial fibrillation: a randomized clinical trial. JAMA. 2013 Nov 20;310(19):2050-60. doi: 10.1001/jama.2013.280521. PMID 24240932
- [Background] Middeldorp ME, Pathak RK, Lau DH, Sanders P. PREVEntion and regReSsive Effect of weight-loss and risk factor modification on Atrial Fibrillation: the REVERSE-AF study-Authors' reply. Europace. 2019 Jun 1;21(6):990-991. doi: 10.1093/europace/euz050. No abstract available. PMID 30887044
- [Background] Yaeger A, Cash NR, Parham T, Frankel DS, Deo R, Schaller RD, Santangeli P, Nazarian S, Supple GE, Arkles J, Riley MP, Garcia FC, Lin D, Epstein AE, Callans DJ, Marchlinski FE, Kolansky DM, Mora JI, Amaro A, Schwab R, Pack A, Dixit S. A Nurse-Led Limited Risk Factor Modification Program to Address Obesity and Obstructive Sleep Apnea in Atrial Fibrillation Patients. J Am Heart Assoc. 2018 Dec 4;7(23):e010414. doi: 10.1161/JAHA.118.010414. PMID 30571593
- [Background] Fernando HA, Zibellini J, Harris RA, Seimon RV, Sainsbury A. Effect of Ramadan Fasting on Weight and Body Composition in Healthy Non-Athlete Adults: A Systematic Review and Meta-Analysis. Nutrients. 2019 Feb 24;11(2):478. doi: 10.3390/nu11020478. PMID 30813495
- [Background] Patterson RE, Sears DD. Metabolic Effects of Intermittent Fasting. Annu Rev Nutr. 2017 Aug 21;37:371-393. doi: 10.1146/annurev-nutr-071816-064634. Epub 2017 Jul 17. PMID 28715993
- [Background] Hussin NM, Shahar S, Teng NI, Ngah WZ, Das SK. Efficacy of fasting and calorie restriction (FCR) on mood and depression among ageing men. J Nutr Health Aging. 2013;17(8):674-80. doi: 10.1007/s12603-013-0344-9. PMID 24097021
- [Background] Teng NI, Shahar S, Manaf ZA, Das SK, Taha CS, Ngah WZ. Efficacy of fasting calorie restriction on quality of life among aging men. Physiol Behav. 2011 Oct 24;104(5):1059-64. doi: 10.1016/j.physbeh.2011.07.007. Epub 2011 Jul 18. PMID 21781980